CLINICAL TRIAL: NCT03590080
Title: Blood Pressure Profile and NT-proBNP Dynamics in Response to Intravenous Methylprednisolone Pulse Therapy of Severe Graves' Orbitopathy
Brief Title: Impact of Intravenous Methylprednisolone Treatment on Blood Pressure
Status: Completed | Type: Observational
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Piotr Miskiewicz, MD, PhD, Medical University of Warsaw
Other Study IDs: IVMPHeart
Record Dates: First submitted 2018-06-30; First posted 2018-07-18 (Actual); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Graves Disease; Graves Ophthalmopathy; Hypertension; Blood Pressure; Heart Failure
Keywords: Graves' Disease; Graves' Ophthalmopathy; Hypertension; Blood Pressure; Methylprednisolone; Glucocorticoids
MeSH Terms: conditions — Graves Disease; Graves Ophthalmopathy; Hypertension; Heart Failure | interventions — Methylprednisolone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — All assays were performed in sera obtained from venous blood samples and analysed immediately after blood sampling in The Central Laboratory in the hospital. NT-proBNP was measured using a Flex® Reagent Cartridge and Dimension®EXLTM integrated chemistry system with a LOCI® Module (Siemens HealthCare Diagnostics Ltd., Camberley, UK). The cutoff value of NT - proBNP typical for hemodynamic stress in the left ventricle was defined as ≥125 pg/ml. Measurements of TnI and hs-CRP were made. Analysis of TnI was performed on Siemens Dimension System (ExL LOCI TnI assay). TnI values ≥ 0.056 ng/mL as above the 99th percentile were reported as positive. Measurement of hs-CRP was performed in serum using an immunoturbidimetric method on Cobas 6000 Analyzer (Roche Diagnostics).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- active, moderate-to-severe GO: Each participant received IVMP according to EUGOGO recommendations (cumulative dose of methylprednisolone 4.5 g, treatment duration 12 weeks in single weekly intravenous pulses, first 6 weeks 0.5g of IVMP, next 6 weeks 0.25g of IVMP).
  Interventions: Drug: Methylprednisolone

INTERVENTIONS:
Drug: Methylprednisolone

SUMMARY:
Hypertension is common side effect of Cushing Syndrome (CS): in patients with endogenous CS and those treated with glucocorticosteroids (GCs). The impact of the intravenous GCs therapy on blood pressure (BP) remains unclear. According to the European Group On Graves' Orbitopathy (EUGOGO), patients with active, severely symptomatic and sight-threatening Graves' orbitopathy (GO) should be treated with high dose intravenous methylprednisolone (IVMP) pulses. There are, however, reports of fatal side effects that may be associated with this therapy (e.g.: pulmonary embolism, myocardial infarction, severe cerebrovascular events, acute liver damage and sudden death). For this reason, the cumulative dose of IVMP should not exceed 8 g within each treatment course, and pulses should not be given on consecutive or alternate days, except for the case of dysthyroid optic neuropathy. A consensus on the monitoring of patients during and after IVMP pulse administration is not yet established. What is more, there is lack of paper regarding pattern of blood pressure at various time points during and after ivGCs administration. Thus, the investigators decided to evaluate acute changes of N-terminal pro-brain natriuretic peptide (NT-proBNP) as a marker of hemodynamic stress and to monitor BP before, during and after IVMP pulse administration. All of patients were treated routinely according to EUGOGO recommendations with standard doses of methylprednisolone with standard recommended schedule. Inclusion criterion for the therapy was according to EUGOGO guidelines active, moderate-to-severe and active GO (12 pulses of IVMP 6x0.5g followed by 6x0.25g every week).

DETAILED DESCRIPTION:
Laboratory tests such as NT-proBNP, troponin I (TnI) and high - sensitivity C - reactive protein (hs-CRP) were performed before, 24 h and 48 h after IVMP during the following pulses: 1st, 6th and 12th. Patients underwent echocardiographic examination before 1st and after 12th pulse. 48-hours ambulatory blood pressure monitoring (ABPM) (for 24 hours before and 24 hours after IVMP) was done during the following pulses: 1st, 6th and 12th.

ELIGIBILITY:
Inclusion Criteria:

* active, moderate-to-severe GO according to EUGOGO classification
* euthyroidism
* completion of at least first six IVMP pulses.

Exclusion Criteria:

* cardiovascular morbidity (such as chronic heart failure and/or coronary heart disease)
* uncontrolled hypertension (defined as systolic blood pressure (SBP) more than 140 mmHg and/or diastolic blood pressure (DBP) more than 90 mmHg)
* contraindications to IVMP therapy
* previous GCs treatment in the last 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the clinic for routine treatment of active, moderate-to-severe GO
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2015-12-30 (Actual); Study Completion 2015-12-30 (Actual)

PRIMARY OUTCOMES:
NT-proBNP 1-24h | 24 hours
  Change in value of NT-proBNP from baseline (before administration of methylprednisolone) to 24 hours after first intravenous pulse
NT-proBNP 1-12w | 12 weeks
  Change in value of NT-proBNP from baseline (before administration of methylprednisolone) to the basic NT-proBNP before last pulse with methylprednisolone
48-hour ambulatory blood pressure monitoring (ABPM)- 1 mean BP | 48 hours
  Analysis of changes in mean blood pressure in ABPM between day before methylprednisolone administration and second day after first pulse of methylprednisolone administration
48-hour ambulatory blood pressure monitoring (ABPM)- 12 mean BP | 12 weeks
  Analysis of changes in mean blood pressure in ABPM between day before methylprednisolone administration and second day after 12th pulse of methylprednisolone administration
48-hour ambulatory blood pressure monitoring (ABPM)- 1 max systolic BP | 48 hours
  Analysis of changes in maximal systolic blood pressure in ABPM between day before methylprednisolone administration and second day after first pulse of methylprednisolone administration
48-hour ambulatory blood pressure monitoring (ABPM)- 12 max systolic BP | 48 hours
  Analysis of changes in maximal systolic blood pressure in ABPM between day before methylprednisolone administration and second day after 12th pulse of methylprednisolone administration
echocardiographic examinations - median values of Ejection Fraction (EF) | 12 weeks
  Analysis of change in median values of EF between echocardiographic examinations before first methylprednisolone administration and after last pulse of methylprednisolone

SECONDARY OUTCOMES:
hs-CRP | 24 hours
  Change in value of hs-CRP from baseline (before administration of methylprednisolone) to 24 hours after first intravenous pulse
Biomarker of cardiomyocyte injury - TnI | 24 hours
  Change in value of TnI from baseline (before administration of methylprednisolone) to 24 hours after first intravenous pulse
NT-proBNP 1-48h | 48 hours
  Change in value of NT-proBNP from baseline (before administration of methylprednisolone) to 48 hours after first intravenous pulse

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Miśkiewicz, MD, PhD, Principal Investigator — Department of Endocrinology Medical University of Warsaw

IPD SHARING:
Plan to Share IPD: Yes
The collected data will be shared in a publication. It includes all laboratory results from all points of evaluation, results of 48 - hour ABPM and echocardiographic measurements
Time Frame: The results of the study will be published in 2018